CLINICAL TRIAL: NCT06761625
Title: Changes in Hormonal Profile and Body Mass Index in Women With Polycystic Ovary Syndrome After Probiotic Intake: A 12-week Placebo Controlled and Randomized Clinical Study
Brief Title: Changes in Hormonal Profile and Body Mass Index in Women With Polycystic Ovary Syndrome After Probiotic Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 1/12/2024
Record Dates: First submitted 2024-12-19; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: PCOS
Keywords: PCOS; probiotics; hormones; BMI

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics Intake (Experimental): The probiotic group received SanProbi® Barrier capsules
  Interventions: Dietary Supplement: SanProbi® Barrier capsules
- Placebo Intake (Placebo Comparator): The placebo group received capsules filled mainly with maize starch and maltodextrins.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: SanProbi® Barrier capsules — The probiotic group received SanProbi® Barrier capsules
  Arms: Probiotics Intake
Other: Placebo — The placebo group received capsules filled mainly with maize starch and maltodextrins.
  Arms: Placebo Intake

SUMMARY:
Changes in hormonal profile and body mass index in women with polycystic ovary syndrome were analised after probiotic intake.

DETAILED DESCRIPTION:
50 women with PCOS , diagnosed based on Rotterdam ESHRE criteria,were assigned to two groups - the probiotics one and the placebo one. Women from the probiotics group were given SanProbi® Barrier capsules. They were taking probiotics for 12 weeks. The placebo group received identical-looking capsules filled mainly with maize starch and maltodextrins. The study concentrates on analysing specific hormones before and after the intervention (giving the probiotics or a placebo to the patients). The serum samples were obtained on days 3-5 (early follicular phase) of menstrual cycle. In the laboratory studies, the following hormones were measured before and after 12-week intervention: Testosterone, Androstenedione, 17-hydroxyprogesterone (17(OH)P); follicle stimulating hormone (FSH), luteinising hormone (LH); estradiol (E2), prolactin (PRL), thyroid stimulating hormone (TSH), thyroxine (T4) and sex hormone binding globulin (SHBG). The weight and height were measured before and after 12-week intervention. BMI was also calculated.

ELIGIBILITY:
Inclusion Criteria:

* women with PCOS, diagnosed based on Rotterdam ESHRE criteria

Exclusion Criteria:

* The patients with comorbidities such as diabetes mellitus type I and II, heart diseas-es, liver diseases, hypertension, hypothyroidism should be excluded from the study

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in hormonal profile after probiotics intake | 12 weeks
  The hormones will be measured before and after 12-week intervention: the main outcome measure will be androstenedione, prolactin, 17-hydroxyprogesterone and testosterone levels measured in ng/ml.

SECONDARY OUTCOMES:
Change in FSH and LH levels in women with polycystic ovary syndrome after probiotic intake | 12 weeks
  LH and FSH levels will be measured before and after 12 weeks of probiotics intake. They are measured in mIU/ml
Change in Estradiol levels in women with polycystic ovary syndrome after probiotic intake | 12 weeks
  Estradiol levels will be measured before and after 12 weeks of probiotics intake. They are measured in pg/ml
Changes in TSH levels in women with polycystic ovary syndrome after probiotic intake | 12 weeks
  TSH levels will be measured before and after 12 weeks of probiotics intake. They are measured in μIU/ml
Changes in SHBG in women with polycystic ovary syndrome after probiotic intake | 12 weeks
  SHBG levels will be measured before and after 12 weeks of probiotics intake. They are measured in nmol/l
Changes in DHEA-S levels in women with polycystic ovary syndrome after probiotic intake | 12 weeks
  DHEA-S levels will be measured before and after 12 weeks of probiotics intake. They are measured in μg/dl
Changes in BMI in women with polycystic ovary syndrome after probiotic intake | 12 weeks
  BMI will be measured before and after 12 weeks of probiotics intake. Weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Locations (1):
- Pomeranian Medical University, Szczecin, Poland

IPD SHARING:
Plan to Share IPD: Undecided